CLINICAL TRIAL: NCT01546467
Title: Cognitive Remediation in Early Phase Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other); South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/1788 (REK)
Record Dates: First submitted 2012-01-12; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Psychosis NOS
Keywords: Schizophrenia; Schizoaffective disorder; Psychosis; Early phase; Cognitive remediation; Functional outcome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive remediation (Experimental): 30 hour computer based cognitive remediation integrated in participants current rehabilitation program (school, work, day program)
  Interventions: Behavioral: Cognitive remediation
- Wait list control group (No Intervention): Participant continues in treatment/rehabilitation program as usual until 9 month assessment when participant receives the same cognitive remediation program as the experimental group.

INTERVENTIONS:
Behavioral: Cognitive remediation — Cognitive remediation including feedback from neurocognitive assessment, psychoeducation about cognitive deficits, 30 hours of computer based drill and practise and strategy coaching based cognitive remediation, 1-3 collaborative meetings with cognitive specialist, participant, therapist and teacher, occupational therapist or other therapist (depending on participants rehabilitation situation) to enhance transfer of skills to daily functioning
  Arms: Cognitive remediation

SUMMARY:
The purpose of the study is to investigate the effect of a 30 hour cognitive remediation program for young patients with early phase schizophrenia spectrum disorders on cognitive, clinical and functional outcome measures. The remediation program is integrated with whatever active rehabilitation the participant is currently attending (school, work, day program etc).

ELIGIBILITY:
Inclusion Criteria:

* Early phase schizophrenia, schizoaffective disorder, psychosis NOS
* Less than 5 years since start of adequate treatment for psychotic disorder
* Age between 18-40
* Norwegian speaking (sufficiently to understand and complete assessments)

Exclusion Criteria:

* Traumatic brain injury
* Neurological disorder as determined by medical history
* IQ below 70

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
MATRICS Consensus Cognitive Battery (MCCB) | Change in MCCB performance from baseline to 4 months and 9 months
  Included in the MCCB are measures of the following cognitive domains: Speed of Processing, Attention, Working memory, Verbal learning, Visual Learning, Reasoning and problem solving and Social Cognition. In addition the following tests are included: HVLT-R and BVMT-R delayed recall to measure memory, TMTB (Halstead Reitan) and Color Word Inteference Test (D-KEFS) to measure executive functioning), Digit span (WAIS-III)to measure working memory, Grooved Pegboard (Halstead Reitan) to measure motor function.
UCSD Performance Based Skilled Assessment Brief Version (UPSA-B) | Change in UPSA-B performance from baseline to 4 months and 9 months
Cognitive Assessment Interview (CAI) | Change in CAI scores from baseline to 4 months and 9 months
Social Functioning Scale (SFS) | Change in SFS scores from baseline to 4 months and 9 months

SECONDARY OUTCOMES:
Calgary Depression Scale | Change in CDS scores from baseline to 4 months and 9 months
Global Assessment of Function (GAF)- split version | Change in GAF scores from baseline to 4 months and 9 months
event related fMRI | Change in BOLD fMRI signal from baseline to 4 months
  Event-related fMRI will be performed to measure neuronal activity during a spatial working memory tasks and an executive planning task. All fMRI data will be collected on Ullevål's 3 T General Electric Sigma HDx scanner.
Rosenberg Self-Esteem Scale (RSES) | Change in RSES scores from baseline to 4 months and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Torill Ueland, PhD, Principal Investigator — Psychosis Research Unit, Division of Mental Health and Addiction, Oslo University Hospital
Locations (1):
- Psychosis Research Unit, Division of Mental Health and Addiction, Oslo University Hospital., Oslo, Norway